CLINICAL TRIAL: NCT07238491
Title: Impact of Virtual Reality on Flexibility, Muscle Strength and Gait Parameters in Young Adults With Hamstring Shortening: A Randomized Controlled Trial
Brief Title: Virtual Reality in Young Adults With Hamstring Shortening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11328
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Hamstring Muscle Tightness
Keywords: virtual reality; Hamstring tightness; flexibility; Muscle strength; gait parameters; young adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Virtual reality group) (Experimental): Participants will receive virtual reality (VR) in addition to the traditional physical therapy program 2 times/week for 5 weeks.
  Interventions: Device: Virtual reality; Other: Traditional physical therapy programme
- Group B (control group) (Active Comparator): Participants will receive a traditional physical therapy program only, 2 times per week for 5 weeks.
  Interventions: Other: Traditional physical therapy programme

INTERVENTIONS:
Device: Virtual reality — A five-minute warm-up, thirty minutes of intervention training, and a five-minute cool-down will all be included in each session. Five minutes of stretching and walking were part of the warm-up. Every participant will play five sports games (running, cool-running, catching gift, football, skate) during each session. These gamed can help teenagers to improve their physical strength, endurance, balance, and coordination. Every game lasted Five minutes.
  Arms: Group A (Virtual reality group)
Other: Traditional physical therapy programme — The exercise programme includes farmer walks, squats, calf raises, stretching exercises, and strengthening activities. The exercises will be performed in one or two sets of 15-20 repetitions, with a 60-second rest in between. The sets, repetitions, and loads will be increased as the participants advance, up to three sets of 60 repetitions for a perceived effort of 70%-80% of 1RM

SUMMARY:
Tightness of hamstring muscle is known as a reduction in range of motion accompanied by a sensation of restriction in the posterior aspect of thigh. Numerous reasons can cause it, such as genetic susceptibility, compensatory tightness due to persistent abnormalities, and muscular strain. Tight hamstrings cause a small amount of knee flexion during exercise and require comparatively high quadriceps efforts to offset the hamstrings' passive resistance. This could result in knee joint pain that affects gait and raise the reaction forces at the patellofemoral joint.

ELIGIBILITY:
Inclusion Criteria:

* Participants with tightness of hamstring muscle with the degree of flexion for knee joint more than 20° throughout active knee extension (AKE) test.
* Their age between 18 and 30 years.
* BMI less than 30 kg/ m2 .
* Sedentary lifestyle that includes sitting on the chair for long period of time for minimum 6 hours per day, 5 days/week for 6 months minimally.
* Participants who did not engaged in a physiotherapy programs in the previous 6 months.
* Absence of fractures, injuries or medications (such as analgesics or muscle relaxants) that may affect the results of the study.

Exclusion Criteria:

* Any neurological diseases (such as; severe disc prolapse and radiating pain).
* Injury of hamstring in the previous 2 years.
* History of knee injury.
* Fracture in lower extremity or the spine.
* Surgery in the spine.
* Unequal leg length > 2cm.
* Congenital deformity.
* Orthopedic disorders such as patellofemoral pain syndrome, musculoskeletal pain, psychiatric problem.
* Any systemic disease, hearing or visual deficits, cognitive, or cardiovascular complications, and pregnancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 5 weeks
  Microfit hand-held dynamometer (HHD) will be used for assessment of hamstring muscle strength. Each participant will lie prone on a standard treatment table. In this position, the participant will be instructed to bend their knee to 90° of knee flexion, where the Microfet 2 MMT-Wireless HHD will be placed on the lower leg, and a downward force toward the table will be held for 5s while the participant resists the downward force. The participant will be instructed to use their maximum effort. It will be performed three times, and an average will be recorded.

SECONDARY OUTCOMES:
Active Knee Extension (AKE) Test | 5 weeks
  A typical, double-arm, plastic goniometer with an arm length of 31.75 cm will be used to measure the AKE angle. With the stationary arm over the thigh and directed to the greater trochanter, and the moving arm over the leg and directed to the lateral malleolus, the goniometer's axis will be fixed over the lateral epicondyle of the femur. The participant will be asked to fully extend the knee of the dominant leg while relaxing their foot. To measure the AKE angle, which is the degree of knee flexion from the last knee extension, they will maintain this position for five seconds.
Step length | 5 weeks
  A GAITRite® electronic walkway system, which includes a walkway with overall measurements of 90 cm × 7 m × 3.2 mm, will be used to assess gait metrics. A 9 m × 4 m laboratory space that is protected from light and noise will be used for the examination of step length. First, participants will be instructed to stand at the start line in an orthostatic position to adopt the start position. Following that, participants will be told to walk along the GAITRite® system's walkway at their own pace, pausing at the goal line.
Stride length | 5 weeks
  A GAITRite® electronic walkway system, which includes a walkway with overall measurements of 90 cm × 7 m × 3.2 mm, will be used to assess gait metrics. A 9 m × 4 m laboratory space that is protected from light and noise will be used for the examination of velocity. First, participants will be instructed to stand at the start line in an orthostatic position to adopt the start position. Following that, participants will be told to walk along the GAITRite® system's walkway at their own pace, pausing at the goal line.
Cadence | 5 weeks
  A GAITRite® electronic walkway system, which includes a walkway with overall measurements of 90 cm × 7 m × 3.2 mm, will be used to assess gait metrics. A 9 m × 4 m laboratory space that is protected from light and noise will be used for the examination of cadence. First, participants will be instructed to stand at the start line in an orthostatic position to adopt the start position. Following that, participants will be told to walk along the GAITRite® system's walkway at their own pace, pausing at the goal line.
Velocity | 5 weeks
  A GAITRite® electronic walkway system, which includes a walkway with overall measurements of 90 cm × 7 m × 3.2 mm, will be used to assess gait metrics. A 9 m × 4 m laboratory space that is protected from light and noise will be used for the examination of velocity. First, participants will be instructed to stand at the start line in an orthostatic position to adopt the start position. Following that, participants will be told to walk along the GAITRite® system's walkway at their own pace, pausing at the goal line.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol